CLINICAL TRIAL: NCT03599934
Title: The Effect of Lifestyle-integrated Functional Exercise Plus a Home Safety Visit on Reducing Falls in Community Older Fallers: a Randomized Controlled Trial
Brief Title: Effect of Home Exercise on Reducing Falls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017.400
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Fall
Keywords: Elderly; Exercise; Fall; Home safety
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LiFE training and home safety assessment (Experimental): The participants will receive Lifestyle Integrated Functional Exercise Program and Home safety assessment
  Interventions: Other: Lifestyle integrated functional exercise program; Other: Home safety assessment
- Control group (No Intervention): The control group will continue their usual daily routine.

INTERVENTIONS:
Other: Lifestyle integrated functional exercise program — Lifestyle-integrated exercise training targeting to improve strength and balance. Strategy to embed the exercise in the daily activity would also be taught so that the life exercise can be performed at any time of the day. The exercise would be taught in 6 home visits over 6-months.
  Arms: LiFE training and home safety assessment
Other: Home safety assessment — Home safety assessment and modification that targets to reduce environmental risk factors of falls.
  Arms: LiFE training and home safety assessment

SUMMARY:
This proposed randomized controlled trial aims to study the long-term compliance of the LiFE program and its combined effects with a home safety visit on fall prevention in community-dwelling older fallers.

DETAILED DESCRIPTION:
This will be a single-blinded randomized controlled trial. The subjects will be randomly assigned to the LiFE exercise plus home safety assessment group, or the control group by a computer program operated by an independent researcher. This study conforms to the ethical principles of the World Medical Association Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or older
* able to ambulate with a Functional Ambulation Category (FAC) score ≥ 3
* able to walk for ≥ 10 meters
* history of falls in the past 12 months
* living in the community
* without MCI or dementia according to the 5-minute Montreal Cognitive assessment
* have a moderate fall risk or above as assessed by the Physiological Profile Assessment
* able to understand Chinese.

Exclusion Criteria:

* blindness
* diagnosis of mental disorders (e.g., severe depression, schizophrenia)
* any contraindications to exercise (e.g. unstable angina).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Fall | 1.5 years
  Prospective fall data will be collected through telephone follow-up for 1.5 year

SECONDARY OUTCOMES:
Handgrip strength | Baseline and follow-up assessment at 6-month
  Hand grip strength will be assessed by handheld dynamometer
Functional lower body strength | Baseline and follow-up assessment at 6-month
  Five-time sit-to-stand test will be used to assess lower body strength
Single leg standing balance | Baseline and follow-up assessment at 6-month
  Single leg standing balance of both legs will be assessed
10-meter walk test | Baseline and follow-up assessment at 6-month
  The usual walking speed on a 10-meter walkway
Timed-up and Go test | Baseline and follow-up assessment at 6-month
  The time required to stand up from a chair, walk 3-m, return, and sit down, in comfortable speed
Timed-up and Go test with dual-task | Baseline and follow-up assessment at 6-month
  The timed-up and Go test would be tested while asking the participants to do serial-3-subtraction
Montreal Cognitive Assessment 5-minute protocol | Baseline and follow-up assessment at 6-month
  A standardized cognitive test
Activity level | Baseline and follow-up assessment at 6-month
  Selected participants will be asked to wear an activity tracker for 7 days to examine their activity level
Fall risk | Baseline and follow-up assessment at 6-month
  Physiological Profile Assessment (PPA) will be used to assess fall risk

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kwok, MD, Principal Investigator — The Chinese University of Hong Kong Jockey Club Centre for Osteoporosis Care and Control
Locations (2):
- Hong Kong (2):
  - The Chinese University of Hong Kong Jockey Club Centre of Osteoporosis Care and Control, Hong Kong
  - The Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided